CLINICAL TRIAL: NCT04222231
Title: Metabolic Effects of a New Resistance Training in Individuals With Type 2 Diabetes
Brief Title: RESIST! Blood-flow Restriction Resistance Training for Improving Insulin Sensitivity in Type 2 Diabetes
Acronym: RESIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: German Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DDZ_Resist
Record Dates: First submitted 2019-12-10; First posted 2020-01-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes
Keywords: Insulin sensitivity; Blood flow restriction training; Muscle hypertrophy; Muscle Strength; Hypoxia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood-flow restriction resistance training (Experimental): Resistance training with low loads (15-30% RM) in combination with a brief occlusion of venous blood flow using a tourniquet while exercising.
  Interventions: Other: Blood-flow restriction resistance training
- Classical resistance training (Experimental): Resistance training with high loads (60-80% RM).
  Interventions: Other: Classical resistance training

INTERVENTIONS:
Other: Blood-flow restriction resistance training — Training program: After 10 minutes of warm-up the participant performs three exercises with BFRT for the lower extremities. The intensity is about 15-30% of 1-RM.
  Arms: Blood-flow restriction resistance training
Other: Classical resistance training — Training program: After warm-up the participant performs three exercises for lower body. The intensity is about 60-80% of 1-RM.
  Arms: Classical resistance training

SUMMARY:
The study aims to investigate the metabolic and cardiovascular effects of classical resistance training with high loads and blood-flow restricted training (BFRT) with low loads in individuals with type 2 diabetes over 12 weeks.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is characterized by an increasing insensitivity of muscle, fat and liver cells to the hormone insulin. About 9% of the global population is affected by this condition and mortality risk is twice as high in individuals with diabetes compared to similar-aged people without diabetes.

Muscle is of particular importance for glucose homeostasis, since in healthy people it accounts for 80-90% of postprandial insulin-stimulated glucose disposal. After cellular uptake of glucose by the specialized glucose transporter 4 (GLUT4), glucose is phosphorylated and stored as glycogen. In individuals with obesity or T2D, the capacity for insulin to facilitate glucose uptake and glycogen synthesis is impaired. This reduced response of a given insulin concentration to exert its biological effect is termed insulin resistance. Subsequent diminished insulin secretion due to β-cell failure results in fasting hyperglycemia and overt diabetes. Importantly, muscle insulin resistance is the initial defect occurring in the development of T2D and precedes the clinical development of the disease by up to 20 years.

Thus, the preservation of skeletal muscle function is essential for people with T2D who have an increased risk of sarcopenia. On the one hand high intensity resistance training (HIT) with 80 % one-repetition maximum (%1-RM) is a well-recognized strategy to improve muscle strength and glycemic control for individuals with T2D, on the other hand elderly or obese people may not be able to tolerate these high loads. Blood flow restriction training (BFRT) with low loads (20-30% 1-RM) has consistently demonstrated comparable effects to HIT and seems to be a promising alternative to increase muscle function.

During the BFRT the muscle becomes hypoxic due to a brief occlusion of venous blood flow using a tourniquet while exercising. Consequently metabolites like lactate, growth hormone (GH) and insulin like growth factor (IGF-1) are released and result in muscle hypertrophy through activating the collagen synthesis and the recruitment of satellite cells. Furthermore cell swelling based on venous blood pooling, reactive hyperemia and metabolite accumulation has been shown to increase protein synthesis by activating the mammalian Target of Rapamycin Complex 1 (mTORC1) pathway. Also, BFRT increases the level of reactive oxygen species (ROS) which may lead to higher glucose uptake during exercise. Last but not least higher threshold motor units (fast twitch fibers) are recruited due to hypoxia and metabolite accumulation.

Although there is a significant inverse relationship between muscle strength and the risk of cardiovascular mortality, cardiovascular adaptations to resistance training are under-explored and poorly understood.

The study therefore aims to investigate the metabolic and cardiovascular effects of BFRT with low loads in individuals with T2D.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age between ≥ 30 and ≤ 69 years
* Individuals with type 2 diabetes
* BMI: 19-40 kg/m²

Exclusion Criteria:

* Acute infections in the last 2 weeks
* Weight fluctuations (> 10% in the last 6 month)
* Therapy with Glitazone, Beta blocker, Insulin
* Malignant cancer
* Heart diseases (angina pectoris, myocardial infarction, acute myocarditis or pericarditis, cardiac wall aneurysms/ stenose, untreated hypotension or hypertension, aortic stenosis, stroke, cardiac insufficiency, NYHA-class ≥II, heart arrhythmia, disturbances of blood circulation in extremities, venous insufficiency, varicose veins)
* Diabetic neuropathy
* Respiratory disease (COPD, Gold grade ≥II)
* Serious heart, kidney or liver disease: - New York Heart Association-Classification (NYHA) stage ≥ II - creatinine ≥ 1.6 mg / dl - Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥ two-fold upper reference value
* Anemia (Hb <12g / l), blood donation in the last 3 month
* Disease of the immune system (leucocytes <5000/μl)
* Application of immunomodulatory agents (Glucocorticoids, Antihistamine, Acetylsalicylic acid)
* Application of antithrombotic agents (Anticoagulant)
* Blood clotting disorders (abnormally levels of thrombocytes [<150.000, >450.000 ± 50 ], Partial thromboplastin time (PTT) [26-36 s ± 5 s], Quick [70-120% ± 10%]) or wound healing
* Thyroid disease (untreated hypothyroidism or hyperthyroidism, treatment with thiamazol)
* Epilepsy
* Application of drugs which can manipulate the thermoregulation (Antipsychotic)
* Rosacea
* Vitamine supplement (with the las 4 weeks)
* Cigarettes (or non-smokers <1 year) alcohol consumption (men> 30 g / d, women> 20 g / d), drug abuse
* Severe psychiatric illness or addiction
* Risk for/ or HIV or Hepatitis B or C
* Shift work or anormal circadian rhythm
* Muscle diseases, orthopedic restrictions
* Hypersensitivity to local anaesthetic
* Pregnancy, lactation
* Metallic and magnetic implants (for example, mechanical heart valves, joint prostheses, clip after vascular surgery, middle and inner ear implants or fresh dental implants)
* Claustrophobia
* Hypohidrosis
* Participation in another intervention study within the last 3 month

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity by blood-flow restriction or classical resistance training | Before and after 12 weeks of training (intervention)
  By using hyperinsulinemic-euglycemic clamp technique, changes in the M-value (mg x kg-1 x min-1) will be measured. The m-value represent the glucose infusion rate at a defined level of hyperinsulinemia during a glucose clamp test. The hyperinsulinemic-euglycemic clamp technique will thus be implicated to assess changes in insulin sensitivity before and after 12 weeks of resistance training.

SECONDARY OUTCOMES:
Changes in skeletal muscle mass by blood-flow restriction or classical resistance training | Before and after 12 weeks of training (intervention)
  Cross-sectional area (cm2) from quadriceps will be measured by MRI imaging technique to evaluate changes in muscle diameter ("hypertrophy") before and after 12 weeks of resistance training.

OTHER OUTCOMES:
Changes in skeletal muscle strength by blood-flow restriction or classical resistance training | Before and after 12 weeks of training (intervention)
  Isometric and submaximal strength tests (kg) will be performed to measure changes in muscle strength before and after 12 weeks of resistance training.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Study Director — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Christiansen D, Eibye KH, Hostrup M, Bangsbo J. Blood flow-restricted training enhances thigh glucose uptake during exercise and muscle antioxidant function in humans. Metabolism. 2019 Sep;98:1-15. doi: 10.1016/j.metabol.2019.06.003. Epub 2019 Jun 12. PMID 31199953
- [Background] Loenneke JP, Fahs CA, Rossow LM, Abe T, Bemben MG. The anabolic benefits of venous blood flow restriction training may be induced by muscle cell swelling. Med Hypotheses. 2012 Jan;78(1):151-4. doi: 10.1016/j.mehy.2011.10.014. Epub 2011 Nov 1. PMID 22051111
- [Background] Abe T, Fujita S, Nakajima T, Sakamaki M, Ozaki H, Ogasawara R, Sugaya M, Kudo M, Kurano M, Yasuda T, Sato Y, Ohshima H, Mukai C, Ishii N. Effects of Low-Intensity Cycle Training with Restricted Leg Blood Flow on Thigh Muscle Volume and VO2MAX in Young Men. J Sports Sci Med. 2010 Sep 1;9(3):452-8. eCollection 2010. PMID 24149640
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Takarada Y, Nakamura Y, Aruga S, Onda T, Miyazaki S, Ishii N. Rapid increase in plasma growth hormone after low-intensity resistance exercise with vascular occlusion. J Appl Physiol (1985). 2000 Jan;88(1):61-5. doi: 10.1152/jappl.2000.88.1.61. PMID 10642363
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Mattocks KT, Jessee MB, Mouser JG, Dankel SJ, Buckner SL, Bell ZW, Owens JG, Abe T, Loenneke JP. The Application of Blood Flow Restriction: Lessons From the Laboratory. Curr Sports Med Rep. 2018 Apr;17(4):129-134. doi: 10.1249/JSR.0000000000000473. PMID 29629973
- [Background] Harreiter J, Roden M. [Diabetes mellitus-Definition, classification, diagnosis, screening and prevention (Update 2019)]. Wien Klin Wochenschr. 2019 May;131(Suppl 1):6-15. doi: 10.1007/s00508-019-1450-4. German. PMID 30980151
- [Background] Pesta DH, Goncalves RLS, Madiraju AK, Strasser B, Sparks LM. Resistance training to improve type 2 diabetes: working toward a prescription for the future. Nutr Metab (Lond). 2017 Mar 2;14:24. doi: 10.1186/s12986-017-0173-7. eCollection 2017. PMID 28270856
- [Background] Centner C, Wiegel P, Gollhofer A, Konig D. Effects of Blood Flow Restriction Training on Muscular Strength and Hypertrophy in Older Individuals: A Systematic Review and Meta-Analysis. Sports Med. 2019 Jan;49(1):95-108. doi: 10.1007/s40279-018-0994-1. PMID 30306467
- See also: Methode — http://www.owensrecoveryscience.com